CLINICAL TRIAL: NCT04330092
Title: Diagnosis of Cow's Milk Protein Allergy Among Infants and Children in Assiut University Children Hospital
Brief Title: Diagnosis of Cow's Milk Protein Allergy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Samir fawzy ali, mohamed samir fawzy ali, Assiut University
Other Study IDs: cow's milk allergy
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will assess the diagnosis of cow's milk protein allergy (CMPA) among infant and children in assiut university children hospital using skin prick test and specific serum IgE as well as their management.

DETAILED DESCRIPTION:
Food allergy is a reproducible specific immune response to exposure to a given food. Cow's milk protein allergy (CMPA) is clinically abnormal reaction to cow's milk protein (CMP) via immune mechanisms triggered by milk protein (Boyce etal.,2010).

According to European academy for allergy and clinical immunology (EAACI) and the world allergy organization (wao) , a hypersensitivity reaction to cow's milk involving the immune system can be called as CMPA. There is difference between CMPA and non-allergic cow's milk intolerance (e.g lactose intolerance) which occurs as a result of lactase deficiency without involvement of the immune system (Venter etal.,2013).

CMPA is categorized into immunoglobulin IgE mediated , non -IgE mediated ,or mixed CMPA (Sicherer etal.,2001).

1.9% to 4.9% prevalence of CMPA among children with a peak in prevalence (2-3%) in the first year of life and prevalence of <1% in children aged >=6 years (koletzko etal.,2012).

ELIGIBILITY:
Inclusion Criteria:

* - Exclusively breast feeding ,breast-fed infants with supplementary foods and non-breast fed infants with supplementary foods who complain from either frequent regurgitation, vomiting,diarrhea,constipation (with/without perianal rash) ,blood in stool or pallor.

Exclusion Criteria:

* : Infant and child with gastrointestinal symptoms due to specific etiology.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: the infant from 1st day to 2 years Exclusively breast feeding ,breast-fed infants with supplementary foods and non-breast fed infants with supplementary foods who complain from either frequent regurgitation, vomiting,diarrhea,constipation (with/without perianal rash) ,blood in stool or pallor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
diagnosis of cow's protein allergy among infants and children from 1st day of life-2 years | baseline
  compare between diagnosis by skin prick test and specific serum IgE

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University, Asyut, Egypt